CLINICAL TRIAL: NCT01005641
Title: Phase II Multicentered Study of Exemestane and Lapatinib in Advanced Hormone-responsive Breast Cancer
Brief Title: ELBA: Exemestane and Lapatinib in Advanced Breast Cancer
Acronym: ELBA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not started for administrative reasons
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Francesco Perrone, NCI Naples
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELBA; EudraCT number: 2008-007946-67
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: advanced breast cancer; hormone-responsive; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): phase II
  Interventions: Drug: exemestane; Drug: lapatinib

INTERVENTIONS:
Drug: exemestane — 25 mg daily
Drug: lapatinib — taken orally, daily, at dose recommended after dose finding part of study

SUMMARY:
Aromatase inhibitors are the standard treatment for hormone responsive advanced breast cancer. The combination of the aromatase inhibitor exemestane with with another breast cancer drug that blocks epidermal growth factor receptor (EGFR) and Erb-2 activity (lapatinib) is being studied for the possibility of improving response to therapy, and delaying resistance to endocrine therapy.

DETAILED DESCRIPTION:
The recommended dose of lapatinib will be determined in the first part of the study. In the second part of the study, patients will receive the recommended dose of lapatinib and exemestane daily, taken orally.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Indication for hormonal therapy (ER and/or PgR positive)
* Stage IV disease
* Female gender
* Postmenopausal status (patients treated with LHRH analogs are eligible for the Phase II part of the study)
* At least one target or non-target lesion according to RECIST criteria
* ECOG Performance Status 0-2
* Adequate bone marrow (neutrophils > or = 1.500/mm³, platelets > or = 100.000/mm³ and hemoglobin > or = 9 g/dl), hepatic (GOT, GPT < 2.5 e bilirubin <1.25 times the value of upper normal limit) and renal (creatinine < 1.25 times the value of upper normal limit) function
* Adequate cardiac function (FEVS > or = 50%)
* Able to take oral medications
* Life expectancy > 3 months
* Signed informed consent

Exclusion Criteria:

* Any previous hormone therapy for metastatic disease
* More than one line of chemotherapy for metastatic disease (first line chemotherapy is permitted)
* Symptomatic cerebral metastases
* Planned concomitant radiation therapy in the first month of therapy (for those patients participating in the dose finding phase of the study)
* Previous therapy with exemestane, including as adjuvant therapy (previous therapy with non-steroidal aromatase inhibitors is permitted)
* Previous or concurrent malignancy in past 5 years (excluding adequately treated basal cel or spinocellular skin cancer and in situ carcinoma of the cervix)
* Treatment with experimental pharmacologic therapy within 4 weeks of enrollment in the study
* Unable or unwilling to provide signed informed consent
* Any concurrent illness that would, in the Investigator's opinion, contraindicate the use of the study drugs.
* Active infection
* Assumption of CYP3A4 inhibitors or inducers (ketoconazole, itraconazole, fluconazole, macrolide antibiotics, antidepressives, calcium-antagonists, cimetidine, carbamazepine, phenytoin, barbiturates, rifampicin e glucocorticoids)
* Pregnancy or lactation
* Unable to comply with follow-up
* Active hepatobiliary disease (with the exception of Gilbert's syndrome, asymptomatic biliary calculi, hepatic metastases or stabile chronic hepatopathy)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
recommended dose of lapatinib given in combination with standard dose of exemestane in patients with advanced hormone-responsive breast cancer | one month after dose selection for each of 3 possible dose levels
proportion of patients free from progression | at 6 months

SECONDARY OUTCOMES:
Treatment related toxicity | every 4 weeks
objective response | at 3 and 6 months
time to progression | at 12 months
overall survival | 18 months
prognostic role of molecular markers and circulating tumor cells | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea de Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Office; Alessandro Morabito, M.D., Principal Investigator — NCI Naples; Nicola Normanno, M.D., Principal Investigator — NCI Naples; Ciro Gallo, M.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (3):
- Italy (3):
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli
  - Ospedale S. Luca ASL SA 3, Vallo della Lucania